CLINICAL TRIAL: NCT05912387
Title: The Effect of Statin Therapy on Bile Acid Physiology and the Microbiome in Primary Sclerosing Cholangitis (PSC): a Multi-omics Study
Brief Title: Statin Therapy in Primary Sclerosing Cholangitis (PSC): a Multi-omics Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha Ranjit Sinha, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 67292
Record Dates: First submitted 2023-06-01; First posted 2023-06-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Primary Sclerosing Cholangitis; Inflammatory Bowel Diseases
Keywords: Statin
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rosuvastatin therapy (Experimental): Participants will receive rosuvastatin for 12 weeks followed by a 2 week washout period prior to the final follow-up visit. All patients will receive the study drug, and will serve as their own control. No participants will receive placebo. Rosuvastatin is FDA approved for treatment of high cholesterol, but its use in this trial is off label.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20 mg tablet once daily by mouth

SUMMARY:
PSC is a liver disease that has no medical cure. Patients with PSC are at a greatly increased risk of cancer and infection. Additionally, many patients require a liver transplant. Progress towards a cure has been severely limited by an incomplete understanding of why patients develop PSC. The investigators aim to close this gap by conducting a pilot human study in patients with PSC, using statin therapy as a model

DETAILED DESCRIPTION:
Database studies have suggested that use of statins is associated with lower mortality in patients with PSC. Statins are also safe, widely used medications for the treatment of high cholesterol. This track record of safety makes repurposing statins for use in PSC an attractive option.

This study will evaluate the impact of bile acid profile and the microbiome. Rosuvastatin induced changes in cell signaling pathways in the body, as well as its impact of bacterial gene expression in the microbiome will be evaluated. The investigators anticipate that this study will provide key insights into the biologic basis of PSC, which may aid in the development of drugs for the treatment of PSC.

This research study will enroll patients with PSC. The study will be conducted in 3 phases: baseline measurements, study period (treatment with rosuvastatin), and follow-up (follow-up after completing statin treatment). All patients will receive the study drug, and no patients will receive placebo treatment. Rosuvastatin is FDA approved for treatment of high cholesterol, but its use in this trial is off label.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, greater than or equal to 18 years of age
* Established diagnosis of PSC, defined by either appropriate cholangiographic findings or supportive liver biopsy plus an established diagnosis of inflammatory bowel disease (IBD - Crohn's disease or ulcerative colitis) per American College of Gastroenterology (ACG) guidelines for the PSC-IBD arm
* Hypercholesterolemia with BMI < 25.0 for the comparison arm

Exclusion Criteria:

* Diagnosis of PSC-autoimmune hepatitis overlap syndrome
* Woman who are pregnant, nursing, or expect to be pregnant
* The presence of any comorbidity known to cause secondary sclerosing cholangitis, including: immunoglobulin G-4 (IgG4), associated cholangitis, recurrent bacterial cholangitis, recurrent pyogenic cholangitis, ischemic cholangiopathy, surgical biliary trauma, cholangiocarcinoma, and portal hypertensive biliopathy
* Diagnosis of a serious medical condition (unless approved in writing by a physician)
* Patients taking statin therapy prior to study initiation
* Patients with known clinically allergy to statin therapy
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 5 times the upper limit of normal
* Bilirubin greater than 3.0 mg/dL
* Recent use of antibiotics (within the last 90 days)
* Concurrent use of any immunosuppressive medications (such as any calcineurin inhibitor, steroids at a dose greater than 10 mg of prednisone-equivalents per day)
* Actively using a fibrate drug
* Actively using a ritonavir containing drug
* Familial hypercholesterolemia or other inherited disorder of lipid metabolism
* Recent myocardial infarction or cerebrovascular accident
* Body mass index > 25.0 for the comparison arm
* Chronic kidney disease stage 5 or end-stage renal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in bile acid (BA) profile: total bile acid | Baseline and week 12
  BA profile of biliary/intestinal aspirate and/or feces in response to statin therapy.
Change in bile acid (BA) profile: secondary bile acids:primary bile acids ratio | Baseline and week 12
  BA profile of biliary/intestinal aspirate and/or feces in response to statin therapy.
Change in bile acid (BA) profile: conjugated:unconjugated BAs ratio | Baseline and week 12
  BA profile of biliary/intestinal aspirate and/or feces in response to statin therapy.
Change in pathogen density in the small intestine | Baseline and week 12
  Measure impact of statin therapy upon pathogen density (ratio of good bacteria to pathogenic bacteria) within the microbial community of the duodenum.
Change in bacterial gene expression profile in the small intestine | Baseline and week 12
  This outcome aims to develop an understanding of the profile of microbial metabolic pathways in the duodenum and changes to the profile in response to statin therapy; gene sequencing with be done using shotgun metagenomics followed by pathway analysis.

SECONDARY OUTCOMES:
Change in bile acid (BA) profile: total bile acid | Baseline, week 4, week 14
  BA profile of biliary/intestinal aspirate and/or feces in response to statin therapy.
Change in bile acid (BA) profile: secondary bile acids:primary bile acids ratio | Baseline, week 4, week 14
  BA profile of biliary/intestinal aspirate and/or feces in response to statin therapy.
Change in bile acid (BA) profile: conjugated:unconjugated BAs ratio | Baseline, week 4, week 14
  BA profile of biliary/intestinal aspirate and/or feces in response to statin therapy.
Change in pathogen density in the small intestine | Baseline, week 4, week 14
  Measure impact of statin therapy upon pathogen density (ratio of good bacteria to pathogenic bacteria) within the microbial community of the duodenum.
Change in bacterial gene expression profile in the small intestine | Baseline, week 4, week 14
  This outcome aims to develop an understanding of the profile of microbial metabolic pathways in the duodenum and changes to the profile in response to statin therapy; gene sequencing with be done using shotgun metagenomics followed by pathway analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha Sinha, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared